CLINICAL TRIAL: NCT06952179
Title: Pericardial Histopathology and COVID-19 Seropositivity in Adult Patients Undergoing First-Time Coronary Artery Bypass Grafting: A Prospective Study
Brief Title: Pericardial Histopathology and COVID-19 Seropositivity
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: kvcsamsun
Record Dates: First submitted 2025-04-29; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Response; COVID-19; Pericardial Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study aims to investigate the association between pericardial histopathologic inflammation grades (acute, chronic, or absent) and COVID-19 seropositivity in adult patients undergoing first-time isolated coronary artery bypass grafting (CABG). Pericardial tissue samples were collected during surgery and evaluated histopathologically, while preoperative COVID-19 serological testing was performed. The primary outcome is to determine whether COVID-19 seropositivity is associated with the severity of pericardial inflammation. Patients with prior cardiac surgery, active COVID-19 infection, systemic inflammatory diseases, chronic immunosuppressive therapy, or malignancy were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Undergoing first-time isolated coronary artery bypass grafting (CABG)
* Availability of pericardial tissue sample for histopathological analysis
* Preoperative COVID-19 serological testing performed
* Written informed consent obtained

Exclusion Criteria:

* Previous history of cardiac surgery (e.g., prior CABG, valve surgery)
* Concomitant cardiac procedures during the same operation (e.g., valve repair, aortic surgery)
* Active COVID-19 infection at the time of surgery (positive PCR test)
* Known autoimmune or systemic inflammatory diseases (e.g., lupus, rheumatoid arthritis)
* Chronic immunosuppressive therapy (e.g., steroids, biologics)
* Known malignancy at the time of surgery

Insufficient or inadequate pericardial tissue sample for histopathological assessment

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included adult patients (≥20 years) undergoing first-time isolated coronary artery bypass grafting (CABG). All patients had available pericardial tissue samples for histopathological evaluation and preoperative COVID-19 serological testing. Patients with prior cardiac surgery, active COVID-19 infection, systemic inflammatory diseases, chronic immunosuppressive therapy, or malignancy were excluded.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pericardial inflammation histopatalogical evaluation | up to 1 year
  prospective evaluation of the relationship between pericardial inflammation grade (0: absent, 1: mild, 2: moderate, 3: severe) and COVID-19 seropositivity in adult patients undergoing first-time coronary artery bypass grafting. The primary outcome of this study is to investigate the association between pericardial inflammation grade, as determined by histopathological evaluation (categorized as acute, chronic, or absent inflammation), and COVID-19 seropositivity in adult patients undergoing first-time coronary artery bypass grafting.

CONTACTS AND LOCATIONS:
Overall Officials: emrah ereren, Study Chair — samsun university Faculty of medicine
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)